CLINICAL TRIAL: NCT05569356
Title: Biomarkers of Inflammation and Autoimmunity: Diagnostic Contribution, Prognosis and Physiopathological Aspects in Arrhythmogenic Cardiomyopathy.
Brief Title: Diagnostic Contribution, Prognosis and Physiopathological Aspects in Arrhythmogenic Cardiomyopathy. (ACORE)
Acronym: ACORE
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210985; 2022-A00283-40 (Other: ANSM)
Record Dates: First submitted 2022-09-14; First posted 2022-10-06 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-03

CONDITIONS: Arrhythmogenic Cardiomyopathy
Keywords: Arrhythmogenic Cardiomyopathy; Inflammatory biomarkers; Autoantibodies
MeSH Terms: interventions — Longitudinal Studies; Retrospective Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, Serum, PBMC, pericardial fluid, myocarditis biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arrhythmogenic Right Ventricular Cardiomyopathy (Prospective)
  Interventions: Biological: Prospective
- Arrhythmogenic Right Ventricular Cardiomyopathy (Retrospective)
  Interventions: Other: Retrospective

INTERVENTIONS:
Biological: Prospective — -Additional blood samples -Myocarditis biopsy sample (routine care) -Additional pericardial fluid sample (routine care)
  Groups: Arrhythmogenic Right Ventricular Cardiomyopathy (Prospective)
Other: Retrospective — None (only data collection)
  Groups: Arrhythmogenic Right Ventricular Cardiomyopathy (Retrospective)

SUMMARY:
This study aims to identify novel inflammatory biomarkers in AC, whether in circulating blood, in situ or as imaging biomarkers to better understand the pathophysiology of the disease and then to determine contribution to the clinical management of patients.

DETAILED DESCRIPTION:
The treatment of AC remains based on palliative measures aimed at treating the consequences of the disease: antiarrhythmic treatments, defibrillator, treatments for heart failure. The identification of new biomarkers, in particular circulating ones, would make it possible to open pathophysiology avenues which, in the long term, could lead to therapies targeted to autoimmunity or inflammation.

Many scientific and medical questions remain unanswered and require precise databases on the diagnostic and prognostic evaluation of this pathology.

The objective of this study is to identify novel inflammatory biomarkers in patients with AC by studying the autoimmunity, inflammatory, and immunological profiles through blood samples and myocardial biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient (age ≥ 18 years old)
2. Patient with a probable or confirmed diagnosis of cardiomyopathy according to the diagnostic criteria of the international task force
3. Patient carrying a pathogenic mutation responsible for cardiomyopathy
4. Patient informed individually of the research

Exclusion Criteria:

1. Patients under curatorship/guardianship
2. Pregnant women
3. Patients who expressed their opposition to participate in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with clinical or preclinical Arrhythmogenic Cardiomyopathy (carrier of risk mutation). The retrospective patients will be informed by mail and the prospective patients will be informed during their routine care visit, both using the opt-out approach.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-10-20 (Estimated); Primary Completion 2032-10-20 (Estimated); Study Completion 2032-10-20 (Estimated)

PRIMARY OUTCOMES:
Measure the correlation between the autoimmunity, inflammatory, and immunological profiles through biomarkers found in blood samples, myocardial biopsies, mass imaging cytometry, and cardiac imaging in patients with Arrhythmogenic Cardiomyopathy (AC) | 10 years

SECONDARY OUTCOMES:
Measure the correlation between circulating biomarkers and the severity of the phenotype determined by the severity of AC and multi-modality imaging | 10 years
Measure the correlation between imaging biomarkers and electrocardiogram (ECG) parameters (presence of repolarization and depolarization abnormalities) | 10 years
Measure the changes in inflammatory biomarkers in serum and cardiac imaging over time | 10 years
Demonstrate a correlation between circulating and imaging biomarkers and the link between the extent of fibro-adipose infiltrates and the ventricular strain | 10 years
Measure the correlation between circulating and imaging biomarker values and electro-anatomical mapping data | 10 years
Screening for cardiotropic virus in pericardial fluid and circulating blood sampled in routine care during epicardial ablation by PCR | 10 years
Measure the correlation between the presence of a pathogenic or common genetic variant and serum/imaging biomarkers. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Estelle GANDJBAKHCH, Dr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Institut de Cardiologie de la Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission Nationale de l'Informatique et des Libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal